CLINICAL TRIAL: NCT03118713
Title: A Phase 4, Randomized, Open-label, Active-controlled, Multicenter Study to Evaluate the Renal Protective Effect (UACR), Efficacy and Safety of Ipragliflozin in Type 2 Diabetes Mellitus Patients With Albuminuria
Brief Title: A Study to Evaluate the Renal Protective Effect (Urine Albumin-to-Creatinine Ratio (UACR)), Efficacy and Safety of Ipragliflozin in Type 2 Diabetes Mellitus Patients With Albuminuria
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision due to enrollment challenges
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1941-MA-3122-KR
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Metformin; Ipragliflozin; Type 2 Diabetes Mellitus; ASP1941; Glimepiride
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; ipragliflozin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ipragliflozin and metformin (Experimental): Subjects will receive daily dosage of ipragliflozin and metformin as single tablets
  Interventions: Drug: metformin; Drug: ipragliflozin
- glimepiride and metformin (Experimental): Subjects will receive daily dosage of glimepiride and metformin as single tablets
  Interventions: Drug: metformin; Drug: glimepiride

INTERVENTIONS:
Drug: metformin — oral
  Other Names: Fortamet; Riomet; Glucophage; Diabex XR; Glumetza; Diabex; Glucophage XR
Drug: ipragliflozin — oral
  Other Names: ASP1941; Suglat
  Arms: ipragliflozin and metformin
Drug: glimepiride — oral
  Other Names: Amaryl
  Arms: glimepiride and metformin

SUMMARY:
The primary purpose of this study is to assess the renal protective effect of ipragliflozin in combination with metformin on the percent change of UACR from baseline to 24 weeks against glimepiride in combination with metformin in type 2 diabetes mellitus patients with albuminuria. The secondary purpose of this study is to assess the efficacy, safety and impact on quality of life (QoL) of ipragliflozin in combination with metformin against glimepiride in combination with metformin in type 2 diabetes mellitus patients with albuminuria.

DETAILED DESCRIPTION:
This is a multicenter study that will compare ipragliflozin/metformin with glimepiride/metformin in the treatment of type 2 diabetes mellitus (T2DM) with albuminuria.

The study will include screening and 24-week treatment period. Subjects entering the study have been on a stable dose of at least 1000 mg/day metformin monotherapy for at least 8 weeks (56 days) prior to Visit 1. For randomization, subject will be stratified by the site and the administration of renin-angiotensin system inhibitors (angiotensin receptor blockers and/or angiotensin-converting-enzyme inhibitors) at Visit 2. Subjects will be centrally randomized to either ipragliflozin/metformin group or glimepiride/metformin group and receive 24-week treatment by each group

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria assessed at Visit 1:

* Subject who is outpatient.
* Subject who has been diagnosed with type 2 diabetes mellitus.
* Subject who has been on a stable dose of at least 1000 mg/day metformin monotherapy for at least 8 weeks (56 days) prior to Visit 1.
* Subject who has an HbA1C value between 7.0% and 9.0% at Visit 1.
* Subject who has a urinary albumin/creatinine ratio greater than or equal to 30 mg/g at Visit 1.
* Subject who has eGFR greater than or equal to 45 mL/min/1.73 m^2.
* Subject is on stable diet and exercise program for at least 8 weeks (56 days) prior to Visit 1.

Inclusion Criterion assessed at Visit 2:

* Subject who has a urinary albumin/creatinine ratio greater than or equal to 30 mg/g at Visit 2.

Exclusion Criteria:

* Subject who has been diagnosed with type 1 diabetes mellitus.
* Subject who started or has changed the types and/or dosage of Renin Angiotensin System (RAS) inhibitors (Angiotensin II Receptor Blockers (ARBs), ACE inhibitors) within 12 weeks prior to Visit 1.
* Subject who has been treated with Sodium-Glucose Cotransporter-2 (SGLT-2) inhibitors within 12 weeks prior to Visit 1.
* Subject who has a history of clinically significant renal disease(s) (other than diabetic nephropathy) such as renovascular occlusive disease, nephrectomy, or renal transplant.
* Subject who has a diabetic ketoacidosis, or history of diabetic ketoacidosis.
* Subject with diabetic coma or precoma.
* Subject with severe infection, serious trauma, or perioperative subject at Visit 1
* Subject who has a history of hypersensitivity to ipragliflozin or glimepiride or other SGLT-2 inhibitors or sulfonylureas.
* Subject has Aspartate Aminotransferase (GOT) (AST) or Alanine Aminotransferase (GPT) (ALT) value exceeding 3 times of upper limit of the normal range, or total bilirubin value exceeding 3 times of upper limit of the normal range at Visit 1.
* Subject has progressive proliferative diabetic retinopathy.
* Subject has a symptomatic urinary tract infection or genital infection at Visit 1.
* Subject has uncontrollable psychiatric disorder(s) with medication.
* Subject abuses drug or alcohol at Visit 1.
* Subject has lactic acidosis or has history of lactic acidosis.
* Subject who has been known to have Hepatitis B, Hepatitis C or Positive Human immunodeficiency virus (HIV).
* Subject is unable or unwilling to adhere to any of the protocol requirements such as hospital visits and dose instruction specified in this study.
* Subject with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
* Subject has participated in another interventional study with study drugs within 12 weeks prior to obtaining written informed consent.
* Subject has a clinical condition which would not allow safe conduct of the study.

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
The percentage of change of Urine Albumin-to-Creatinine Ratio (UACR) | Baseline up to 24 weeks
  Early morning urinary sample will be collected for the test

SECONDARY OUTCOMES:
The percentage of patients whose UACR level is normalized or improved more than 50% | Baseline up to 24 weeks
  Early morning urinary sample will be collected for the test
Change from baseline in Estimated glomerular filtration rate (e-GFR) | Baseline up to 24 weeks
  Test parameter e-GFR shall be measured at the local laboratory
Change from baseline in Hemoglobin A1c (HbA1c) | Baseline up to 24 weeks
  Test parameter HbA1c shall be measured at the local laboratory
Change from baseline in Fasting Plasma Glucose (FPG) | Baseline up to 24 weeks
  Test parameter FPG shall be measured at the local laboratory
Change from baseline in body weight | Baseline up to 24 weeks
  Body Weight shall be measured by the same scale for the clinical trial period
Change from baseline in blood pressure | Baseline up to 24 weeks
  Blood pressure will be measured two times with 1-2 minutes interval by the same arm and procedure during the study
Change from baseline in Uric Acid | Baseline up to 24 weeks
  Test parameter Uric Acid shall be measured at the local laboratory
Change from baseline in health status as measured through EuroQol 5 Dimension 5 Level Health State Utility Index (EQ-5D-5L) questionnaire | Baseline up to 24 weeks
  The EQ-5D-5L Questionnaire consists of 5 domains: mobility, self-care, usual activities, pain/discomfort, anxiety/depression
Change from baseline in health status as measured through EuroQol-Visual Analogue Scale (EQ VAS) questionnaire | Baseline up to 24 weeks
  The EQ VAS measures the score (0 to 100) of change from baseline to 24 weeks
Change from baseline in Quality of Life as measured through Audit of Diabetes-Dependent Quality of Life-19 (ADDQoL-19) questionnaire | Baseline up to 24 weeks
  Quality of Life will be assessed through ADDQoL-19. Patients will be asked to complete the questionnaires at visit 2 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Korea, Inc.
Locations (8):
- South Korea (8):
  - Site 13, Busan
  - Site 02, Deagu
  - Site 11, Guri-si
  - Site 01, Seoul
  - Site 05, Seoul
  - Site 07, Seoul
  - Site 09, Seoul
  - Site 12, Suwon

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=359